CLINICAL TRIAL: NCT00459654
Title: A Phase II Randomised, Placebo-controlled, Multicentre Study in Prostate Cancer Patients With Painful Bone Metastases to Evaluate the Efficacy of Repeated Radium-223 Injections
Brief Title: A Placebo-controlled Phase II Study of Bone-targeted Radium-223 in Symptomatic Hormone-refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15280; BC1-02 (Other: Algeta ASA)
Record Dates: First submitted 2007-04-11; First posted 2007-04-12 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Prostate Cancer; Neoplasm Metastasis
Keywords: HRPC; Recurrent Prostate Cancer; Metastatic Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — radium Ra 223 dichloride; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radium-223 dichloride (Xofigo, BAY88-8223) (Experimental): Each subject receives local filed external beam radiotherapy (EBR) and repeated injections of the investigational drug radium-223 (EBR+Radium-223)
  Interventions: Drug: Radium-223 dichloride (BAY88-8223)
- Saline (Placebo Comparator): Each subject receives local filed external beam radiotherapy (EBR) and repeated injections of saline (EBR+placebo)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Radium-223 dichloride (BAY88-8223) — Four Radium-223 injections were given at 4-weekly intervals starting after the first fraction of EBR.
  Arms: Radium-223 dichloride (Xofigo, BAY88-8223)
Drug: Saline — Four Saline injections were given at 4-weekly intervals starting after the first fraction of EBR.
  Arms: Saline

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the investigational radioisotope Radium-223 in treatment of men with prostate cancer and bone metastases that no longer respond to hormonal treatment.

DETAILED DESCRIPTION:
Primary objective:

To study the biological effectiveness of radium-223 therapy measured as:

* Time to occurrence of skeletal-related events(SREs)
* Change in bone-specific alkaline phosphatase (bone-ALP) levels

Secondary objectives:

To study the efficacy of radium-223 therapy in terms of:

* Frequency of new SREs
* Proportions of patients with an SRE
* Proportions of patients with SRE at different time points
* Changes of biochemical markers of bone turnover
* Treatment response with regard to pain and analgesic use(termed "Palliative effect" in study protocol)
* Quality of life assessment
* Overall survival To study the safety of the repeated radium-223 regimen Total Enrollment:64 Study start: February 2004

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed adenocarcinoma of the prostate
* Patient has received or is receiving hormonal treatment (orchiectomy, polyoestradiol phosphate, or gonadotropin-releasing hormone analogue with or without antiandrogen)
* Metastatic disease with positive bone scan within 2 months before treatment with more than one cancer related lesion or with one painful cancer related lesion in the presence of increasing PSA levels as follows: PSA >5 ng/ml, with increases on at least 2 successive occasions at least 2 weeks apart.
* Patient is referred to local field radiotherapy (EBR) for metastatic bone pain. The area to be treated (index site) should match the positive bone scan, local radiation area not exceeding 400 cm2
* ECOG performance status: 0-2
* Life expectancy: at least 3 months
* Age more than 40 years
* Laboratory requirements:

  * Hematology: Neutrophil count ≥1,5 x 109/L Platelet count at least ≥100 x109/L and stable Hemoglobin >100 g/l or 10 g/dL
  * Hepatic function: Bilirubin within normal institutional limits ASAT and ALAT <2,5 times upper limit of normal (ULN)
  * Renal function: Creatinine <1,5 times the ULN (i.e. NCI grade ≤1)
* Patient is willing and able to comply with the protocol, and agrees to return to the hospital for follow-up visits and examinations
* Patient has been fully informed about the study and has signed the informed consent form

Exclusion Criteria:

* Has received an investigational drug in the 4 weeks before or is scheduled to receiving one during the planned treatment period
* Has received chemo-, immunotherapy or external radiotherapy within weeks before study drug administration
* Has started treatment with bisphosphonates within 3 months before administration of study drug.
* Has previously received systemic radiotherapy with strontium, samarium or rhenium
* Change in hormonal therapy within the last 6 weeks before study drug administration
* Other currently active (relapse within the last 3 year) malignancy (except nonmelanoma skin cancer) or known brain, liver, lung, visceral and lymphatic metastases dominating the clinical picture of the patient
* Has received blood transfusion within last month
* Other serious illness or medical condition as follows:

  * any uncontrolled infection
  * heart insufficiency, grade 3 or 4 as specified in NCI-CTC criteria
  * grade 2 or greater motor or sensory neuropathy
  * Crohn's disease or Ulcerative colitis 9) Known non-pathological bone fracture within the last two months

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2004-02; Primary Completion 2006-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Time to occurrence of Skeletal-related Events (SRE) | Up to 12 Month
  SREs are defined as: Increase in pain severity index during the last week; Increase in analgesic consumption; Neurological symptoms secondary to skeletal manifestations of prostate cancer; New pathologic bone fractures (vertebral and non-vertebral); Tumour related orthopaedic surgical intervention; Subsequent external beam radiation to relieve skeletal pain; Use of radioisotopes to relieve new skeletal related symptoms; Use of corticosteroids for skeletal pain, at doses aimed for pain palliation; Use of chemotherapy, bisphosphonates, or hormones, for the treatment of skeletal disease progression
Relative change (%) in bone-ALP levels from baseline to 4 weeks after last injection | Up to 12 Month

SECONDARY OUTCOMES:
Number of SREs per patient | Up to 12 Month
Changes in the levels of biochemical markers of bone formation | Up to 12 Month
Change in Prostate Specific Antigen (PSA) | Up to 12 Month
Change in pain level | Up to 12 Month
Changes in analgesic use during study period | Up to 12 Month
Changes in Edmonton Symptom Assessment Scale (ESAS) from baseline | Up to 12 Month
Overall survival | up to 24 months
Adverse events | up to 24 months
Clinical laboratory tests including haematology, renal and liver function parameters | up to 24 months

CONTACTS AND LOCATIONS:
Locations (3):
- Sweden (2):
  - Linköping
  - Sundsvall
- Nottingham, United Kingdom